CLINICAL TRIAL: NCT02415101
Title: Randomized Clinical Trial Comparing the Timing of Resective Surgery After Neoadjuvant Chemoradiotherapy in Cancer of the Esophagus or Gastric Cardia
Brief Title: Timing of Resective Surgery After Neoadjuvant Chemoradiotherapy in Esophageal Cancer
Acronym: NeoResII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Oslo University Hospital (Other); Lund University Hospital (Other); Sahlgrenska University Hospital (Other); Region Örebro County (Other); University Hospital, Umeå (Other); St. Olavs University Hospital (Unknown); University Hospital, Linkoeping (Other); University Hospital of North Norway (Other); University Hospital Cologne (Unknown)
Responsible Party: Principal Investigator, Magnus Nilsson, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/748-31-3
Record Dates: First submitted 2015-02-22; First posted 2015-04-14 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2024-03

CONDITIONS: Cancer of the Esophagus
Keywords: Adenocarcinoma; Squamous cell carcinoma; Gastroesophageal Junction
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resective surgery after 4-6 weeks (Active Comparator): Resective surgery 4-6 weeks after completed chemoradiotherapy (CRT)
  Interventions: Procedure: Resective surgery
- Resective surgery after 10-12 weeks (Active Comparator): Resective surgery 10-12 weeks after completed chemoradiotherapy (CRT)
  Interventions: Procedure: Resective surgery

INTERVENTIONS:
Procedure: Resective surgery

SUMMARY:
This study compares outcomes with regard to the timing of resective surgery after neoadjuvant chemoradiotherapy (CRT) in cancer of the esophagus or gastric cardia. Patients are randomised to surgery either conventional 4-6 or 10-12 weeks after termination of CRT. The study hypothesis is that a longer delay improves histological response and decreases the risk of postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma or SCC of the esophagus or GEJ Siewert type I and II.
* Tumors should be resectable and without distant metastasis, as assessed after completed CRT.
* Patients with performance status 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale at the pre CRT evaluation and judges to be fit for surgery at the pre and post CRT evaluations.
* Pre CRT tumor stage: T1N1-3M0, T2N0-3M0, T3N0-3,M0, T4aN0-3,M0
* Written informed consent
* Completed at least 80% of the planned chemotherapy and at least 90% of the prescribed radiotherapy dose within the neoadjuvant CRT schedule according to protocol within a period of <36 days.

Exclusion Criteria:

* Concomitant malignant diagnosis (excluding non-melanoma skin cancer) <5 years since current cancer diagnosis.
* Ongoing antitumoral treatment irrespective of time since diagnosis of earlier malignancy.
* Patients being unable to comply with the protocol for reasons of language or cognitive function.
* Tumor stage T1N0, T4bNX or TXNXM1.
* Carcinoma of the upper third of the esophagus (i.e. cervical and uppermost thoracic) for simplicity here defined as upper border of tumor above 22 cm from incisors at endoscopy.
* Clear radiological signs of tumor progression during CRT on CT-scan after completion of CRT. PET is not used in this decision as FDG-activity often increase due to radiotherapy induced inflammation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Complete histological response proportion, using the Chirieac grading system. | analysis is completed 4 weeks after surgery

SECONDARY OUTCOMES:
Overall primary tumor treatment response defined as complete histological response (Chirieac 0) and partial histological response (Chirieac 1 and 2) together. | analysis is completed 4 weeks after surgery
ypN tumor status, classified as ypN0 to ypN3. | analysis is completed 4 weeks after surgery
5 year survival by intention to treat and per protocol analyses in each study arm. | 5 years
Proportion of disease free patients after 5 years by intention to treat and per protocol analyses in each study arm. | 5 years
R0 resection rate in each study arm. | analysis is completed 4 weeks after surgery
Resectability rate in each study arm. | 4-6 or 10-12 weeks after completed CRT
Safety and toxicity (only grade 3-5 toxicity will be reported) ety and toxicity (only grade 3-5 toxicity will be reported) | 4-6 or 10-12 weeks after completed CRT
  According to Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
Postoperative complications in each study arm. | 30 days after surgery
  Using the classification in the Swedish National Registry for Gastric and Esopgageal Cancer (NREV), including Clavien-Dindo classification.
Health-related quality of life (HRQOL). | 4-6 or 10-12 weeks prior to surgery (at randomization after completed CRT), within a week before surgery, 6 months postoperatively, 12 months postoperatively and then yearly until 5 years of follow-up.
  Validated questionnaires that assess patients functions (physical, emotional, social, role and cognitive function), symptoms (e.g. fatique, pain, nausea/vomiting, appetite, dysphagia, eating difficulties and diarrhea) and global quality of life.
QUALYs at 5 year follow-up in each study arm. | 5 years after surgery
  Quality Adjusted Life Year assesses not only how much longer the treatment will allow the patient to live, but weighs in the quality of life with survival as a composite variable.
Correlation between symptom scores, endoscopy and radiology; and complete histological response. | 4 weeks after surgery
Nutritional status of patients in each study arm. | within a week before the start of CRT, within a week before surgery and 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nilsson, Prof, Principal Investigator — Karolinska University Hospital
Locations (1):
- Department of Surgery Gastrocentrum Karolinska Univeristy Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Nilsson K, Klevebro F, Rouvelas I, Lindblad M, Szabo E, Halldestam I, Smedh U, Wallner B, Johansson J, Johnsen G, Aahlin EK, Johannessen HO, Hjortland GO, Bartella I, Schroder W, Bruns C, Nilsson M. Surgical Morbidity and Mortality From the Multicenter Randomized Controlled NeoRes II Trial: Standard Versus Prolonged Time to Surgery After Neoadjuvant Chemoradiotherapy for Esophageal Cancer. Ann Surg. 2020 Nov;272(5):684-689. doi: 10.1097/SLA.0000000000004340. PMID 32833767